CLINICAL TRIAL: NCT05101759
Title: Impact of Chemotherapeutic Treatments on Functional Autonomy and Quality of Life in Patients Aged 75 Years and Over Treated for Lymphoid Hematological Malignancy
Brief Title: Impact of Chemotherapeutic Treatments in Patients Aged 75 Years and Over Treated for Lymphoid Hematological Malignancy
Acronym: LYMPHOLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/20/0490
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Neoplasm, Plasma Cell; Lymphoma
Keywords: comprehensive geriatric assessment (CGA); quality of life (QoL); autonomy; elderly patients; chemotherapy; immunochemotherapy; lymphoma
MeSH Terms: conditions — Neoplasms, Plasma Cell; Lymphoma | interventions — Geriatric Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Geriatric Follow-up (Comprehensive Geriatric Assessment) (Other): A systematic reassessment of geriatric parameters
  Interventions: Procedure: Comprehensive Geriatric Assessment

INTERVENTIONS:
Procedure: Comprehensive Geriatric Assessment — A systematic reassessment of geriatric parameters will be performed at 3 and 6 months post-inclusion.

SUMMARY:
The aim of the study is to assess the prevalence of functional decline in elderly patients treated with chemotherapy or immunochemotherapy for lymphoid hematologic malignancies. For this purpose, each patient benefits at inclusion (D0) of a standardized gerontological evaluation, and 3 and 6 months post-inclusion.

DETAILED DESCRIPTION:
The aim of this study is to contribute to the improvement of the hematological management of elderly patients. Indeed, the majority of hematological malignancies are diagnosed in subjects aged 65 years and over. Hematologists are therefore increasingly confronted with the complexity of managing elderly patients. The high prevalence of comorbidities and/or geriatric syndromes (cognitive disorders, malnutrition, loss of functional autonomy, etc.) contributes to the great heterogeneity of this population and to the complexity of therapeutic decisions.

The comprehensive geriatric assessment (CGA), recommended by the International Society of of Onco-Geriatrics (SIOG), allows to better understand this heterogeneity and to define an individualized management. Numerous studies have demonstrated the value of the CGA in predicting the risk of treatment toxicity and morbidity in geriatric hematology. However, beyond life expectancy, the maintenance of quality of life and/or functional autonomy represent major parameters to be integrated into the therapeutic decision. These two parameters are not sufficiently taken into account in hematology clinical trials. In the vast majority of these studies, the criteria of interest remain purely hematological (overall survival, toxicity, relapse-free survival, etc.). This approach may even be responsible for an increased risk of toxicity when the chemotherapy protocols proposed to elderly patients are based on the same objectives as those for younger subjects. It therefore seems essential to change the paradigm by integrating major geriatric criteria into the methodology of clinical trials of hematological malignancies in elderly patients.

The main objective of our study is therefore to evaluate the prevalence of functional decline in a population of elderly patients treated with chemotherapy or immuno-chemotherapy for lymphoid hemopathies. For this purpose, each patient benefits at inclusion (D0) of a standardized gerontological evaluation, and 3 and 6 months post-inclusion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 75 years of age or older,
* Lymphoid hemopathies (diffuse large cell B-cell lymphoma (DLBCL), follicular lymphoma, marginal zone lymphoma, Hodgkin's lymphoma and T-cell lymphoma, chronic lymphocytic leukemia (CLL)) or plasma cell and/or lymphoplasmacytic hemopathies (multiple myeloma or Waldenström disease).
* World Health Organization (WHO) performance index 0-3,
* Patients requiring first or second line chemotherapy and/or immunotherapy associated or not to targeted therapy,
* Patients with a life expectancy of more than 3 months,
* Persons affiliated or benefiting from a social insurance,
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* Myeloid hemopathies,
* Patient included in a clinical trial that potentially interferes with the purpose of the study (geriatric interventional study, early drug study),
* Patient under court protection, guardianship or curator

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Functional Decline | 6 months
  Rate of patients with functional decline at 6 months. Functional decline was defined as a loss of 0.5 points or more on the Activities Daily Living scale (ADL) at 6 months compared with inclusion.

SECONDARY OUTCOMES:
Functional performance | 6 months
  A loss of at least 1 point in the Short Physical Performance Battery (SPPB) score
Toxicity assessed according to NCI-CTCAE v5 | 6 months
  Events of Toxicity will be assessed according to NCI-CTCAE v5
Institutionalization | 6 months
  Ratio of institutionalized patients to total patients
Early death | 6 months
  Ratio of the number of patients who died early

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BALARDY, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France, France

IPD SHARING:
Plan to Share IPD: No